CLINICAL TRIAL: NCT02547194
Title: Graft Patency as a Predictor of Health-related Quality of Life in Coronary Artery Bypass Patients.
Brief Title: Graft Patency as a Predictor of Health-related Quality of Life.
Status: Completed | Type: Observational
Sponsor: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Ninos Samano M.D., Cardiothoracic Surgeon, Örebro University, Sweden
Other Study IDs: 167861
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Ischemic Heart Disease; Atherosclerosis
Keywords: coronary artery bypass grafting; saphenous vein; no-touch technique
MeSH Terms: conditions — Myocardial Ischemia; Atherosclerosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No touch vein grafts: The grafts were harvested with there surrounding tissues.
- Conventional vein grafts.: The grafts were stripped from surrounding tissue.

SUMMARY:
The health-related quality of life questionnaire "EQ-5D" has been collected in connection with several interventional and observational studies where the no-touch vein harvesting technique in CABG has been used. The results of the questionnaires will be compiled and reported in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Operated at our department for a coronary artery bypass surgery with either the no-touch harvesting technique of conventional harvesting technique.
2. Completed the EQ-5D questionnaire.
3. Signed and dated consent.

Exclusion Criteria:

1. Substantial missing data from the EQ-5D questionnaire.
2. Unable to comprehend the different inquiries in the questionnaire.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients included in the study have been operated on at the department of Cardiothoracic and Vascular Surgery, Orebro University Hospital, Orebro, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The health-related quality of life. | 5-15 years postoperatively.
  EQ-5D is a generic measure of health. The instrument can be used to measure quality of life change in a population over time and to compare the quality of life among different groups in the population such as different socio-economic groups. EQ-5D is constructed of five dimensions: mobility, care, usual activities, pain / discomfort and anxiety / depression. Each dimension is answered on a three-point scale (none, moderate or severe symptoms). With this instrument, it can theoretically be 243 possible health conditions. Health condition can also be described as an index value between 0 corresponding to death and one equivalent full health. Some negative values corresponding a state worse than death can occur. Moreover consists EQ-5D of a VAS scale (Visual Analogue Scale), a thermometer-like scale, with 0 being the worst possible health status and 100 representing full health.

CONTACTS AND LOCATIONS:
Overall Officials: Ninos Samano, MD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Department for Cardiothoracic and Vascular Surgery, Örebro University Hospital, Örebro, Sweden

REFERENCES:
- [Derived] Samano N, Bodin L, Karlsson J, Geijer H, Arbeus M, Souza D. Graft patency is associated with higher health-related quality of life after coronary artery bypass surgery. Interact Cardiovasc Thorac Surg. 2017 Mar 1;24(3):388-394. doi: 10.1093/icvts/ivw372. PMID 28040753